CLINICAL TRIAL: NCT05970965
Title: Study of Neutrophils During Gingival Inflammation in Children With Down Syndrome/Trisomy 21
Brief Title: Periodontitis and Inflammation in Children With Down Syndrome/Trisomy 21: Study on Biological Samples
Acronym: NT21
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP230786
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Periodontitis; Trisomy 21
Keywords: Down syndrome; Trisomy 21; psychomotor retardation; gingivitis; periodontitis; neutrophils; biological collection
MeSH Terms: conditions — Periodontitis; Down Syndrome; Psychomotor Disorders; Gingivitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Child patient consulting the service (Experimental): * Trisomy 21 patient with gingival inflammation (subgroup 1)
  * Trisomy 21 patient with healthy gingiva on intact periodontium with no history of periodontitis (subgroup 2)
  * Patient with psychomotor retardation with no known repercussions on the orofacial sphere or immunity, presenting gingival inflammation (subgroup 1)
  * Patients with psychomotor retardation and no known repercussions on orofacial health or immunity, presenting gingival health on intact periodontium with no history of gingival inflammation (subgroup 2).
  * Patients with no known general pathology and gingival inflammation (subgroup 3)
  * Patients with no known general pathology and healthy gingiva on intact periodontium with no history of gingival inflammation (subgroup 4)
  Interventions: Procedure: Biological sampling

INTERVENTIONS:
Procedure: Biological sampling — - Saliva and blood sampling

SUMMARY:
Since 2018, the Chicago Classification of Periodontal Diseases and Conditions, has listed Down syndrome (DS)/trisomy 21 (T21) as a systemic disease with periodontal implications. Numerous studies report an increased prevalence and severity of periodontitis in DS/T21 individuals under the age of 35. Approximately 35% of adolescents with DS show early signs of alveolar bone loss. However, very few studies have examined the role of immune deficiency in DS/T21 patients in the pathogenesis of periodontitis. Indeed, periodontitis induced by bacterial plaque is virtually non-existent in the paediatric population, leaving the field to systemically-induced periodontitis.

The investigators hypothesize that specific neutrophil phenotypes in DS/T21 patients are key to explaining the rapid progression to periodontitis.

Investigator's primary objective is to characterize the different oral and blood neutrophil subtypes in DS/T21 children with gingival inflammation.

Investigator's secondary objective is to assess the involvement of different neutrophil subtypes in early periodontitis in children with DS/T21.

DETAILED DESCRIPTION:
It's a cross-sectional, monocenter, prospective, open-label, non-randomized case control study to collect saliva and serum samples as part of the patient's routine care in oral medicine department to form a biological collection.

Patients will be recruited in the oral medicine department of AP-HP Charles Foix hospital (Ivry/Seine) by periodontists in 2 groups (CASES: Group 1 for children with DS/T21 divided into 2 subgroups according the periodontal health, and CONTROLS: Group 2 divided into 4 subgroups according to the systemic and periodontal health) Inclusion period is 12 months. There is no specific follow-up due to the research.

Assessment criteria:

* Primary criteria: Neutrophil subtypes analysis based on co-expression of neutrophil function markers from a panel of 24 markers by flow cytometry.
* Secondary criteria: assessment of neutrophil sub-types present in the patient's saliva and study of the correlation within blood neutrophils, during periodontal health, gingivitis and periodontitis.

ELIGIBILITY:
Inclusion Criteria:

Common to all groups:

* Age: 3 to 12
* Patient affiliated to a social security program, beneficiary not covered by the AME.
* Legal representatives who speak and understand French well enough to be able to read and understand the study information.
* Legal representatives giving written consent for their child's participation in the study.

Specific:

Case Group:

* Trisomy 21 patient with gingival inflammation (subgroup 1)
* Trisomy 21 patient with healthy gingiva on intact periodontium with no history of periodontitis (subgroup 2)

Control Group: child meeting one of these criteria:

* Patient with psychomotor retardation with no known repercussions on the orofacial sphere or immunity, presenting gingival inflammation (subgroup 1)
* Patients with psychomotor retardation and no known repercussions on orofacial health or immunity, presenting gingival health on intact periodontium with no history of gingival inflammation (subgroup 2).
* Patients with no known general pathology and gingival inflammation (subgroup 3)
* Patients with no known general pathology and healthy gingiva on intact periodontium with no history of gingival inflammation (subgroup 4)

Exclusion Criteria:

Common to all groups:

* Patient having received antibiotic prophylaxis, antibiotic therapy or anti-inflammatory treatment in the 3 months prior to inclusion
* Patient included in another interventional research protocol or in a period of exclusion.
* Patient on AME
* Patients with a contraindication to the use of MEOPA:

  * Patients requiring pure oxygen ventilation
  * Intracranial hypertension
  * Unevaluated head trauma
  * New-onset, unexplained neurological abnormalities
  * Pneumothorax
  * Emphysema bubbles
  * Gas embolism
  * Diving accident
  * Abdominal gas distension, occlusion
  * Patient recently treated with ophthalmic gas (SF6, C3F8, C2F6)
  * Known, unsubstituted vitamin B12 deficiency

Specific to Trisomy 21 group:

- Patient with no genetic diagnosis

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Distinction of neutrophil subtypes according to co-expression of markers of neutrophil function among a panel of 24 markers by flow cytometry | 1 year
  purification od neutrophils from blood and saliva Fixation Cell sorting using FACS on a panel of 24 markers

SECONDARY OUTCOMES:
Evaluation of neutrophil subtypes present in saliva and study of a correlation with blood neutrophils during periodontal health and periodontal inflammation (intra individual analysis) | 1 year
  Correlation with previous results

CONTACTS AND LOCATIONS:
Overall Officials: Marjolaine Ms GOSSET, PU-PH, Principal Investigator — APHP
Locations (1):
- Carles-Foix Hospital, Ivry-sur-Seine, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request :
  The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.